CLINICAL TRIAL: NCT00288665
Title: Thrombectomy Before Primary Percutaneous Coronary Intervention for Acute Myocardial Infarction Improves Left Ventricular Function at 3 Months
Brief Title: Thrombectomy and Improvement of Left Ventricular Function in AMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: R&D Cardiologie (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Versie 1.0 d.d. 1-7-2004
Record Dates: First submitted 2006-02-06; First posted 2006-02-08 (Estimated); Last update posted 2006-02-08 (Estimated); Status verified 2006-02

CONDITIONS: Acute Myocardial Infarction; Ventricular Remodeling
Keywords: Myocardial infarction; aspiration; thrombectomy; ventricular remodeling
MeSH Terms: conditions — Ventricular Remodeling; Myocardial Infarction

INTERVENTIONS:
Device: Export catheter (Medtronic)

SUMMARY:
To study the effect of a simple and fast 'modus operandi' by aspiration of thrombus and debris with the Export catheter in an acute occlusion, on microvascular (re)perfusion and late left ventricular remodeling. Subsequently determinating if PCI with primary aspiration as an adjunct is superior to standard PCI. Microvascular (re)perfusion will be assessed with angiographic and electrocardiographic measurements (TIMI frame count, TIMI flow grade, Blush score, ST-T segment measurements). Early and late left ventricular function and infarct size will be measured with serial MRI imaging.

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) has dramatically improved mortality and morbidity in patients suffering an acute ST elevation myocardial infarction. Infarct size reduction, prevention of recurrent infarction and improved wound healing are thought to be the mechanisms responsible for the short and long-term clinical benefit of the procedure. In spite of this, myocardial salvage after PCI is often suboptimal because of distal embolisation of atherothrombotic debris and intense microcirculatory vasoconstriction caused by vasoactive substances released from platelets. This will cause a larger infarcted area with increased early and late left ventricular remodelling. Prevention of debris embolisation is therefore a potentially way to further improve myocardial salvage and thus mortality in patients suffering an acute myocardial infarction.

One approach towards embolisation prevention is intracoronary thrombectomy before PCI. Current thrombectomy devices can be classified as fragmentation/suction devices such as the X-sizer catheter and the AngioJet device and the more simple and less costly suction-only devices such as the Export catheter, the Diver CE aspiration catheter (10) and the Rinspiration system. In trials published so far improved outcome has been shown with endpoints representing myocardial perfusion such as ST-T segment resolution, TIMI flow grade, TIMI frame count and myocardial blush grade. These trials were not powered to show differences in clinical end-points.

White et al (11) showed that the best predictor of survival after initial recovery from myocardial infarction is left ventricular end-systolic volume index (ESVI). Regional and global left ventricular function and morphology can be quantified with high reproducibility by cine magnetic resonance imaging (MRI)(12). The method is safe, non invasive, well validated and is at the moment the standard of reference for left ventricular function assessment. The high reproducibility of the technique allows the detection of between-group differences in LV volumes with relatively few patients. This makes MRI measured left ventricular end systolic volume index a very attractive surrogate end-point for small hypothesis forming clinical trials.

We therefore conducted a randomized trial with MRI assessment of LV volumes to evaluate the effect of intracoronary thrombectomy prior to mechanical reperfusion therapy in AMI on early and late left ventricular remodelling

ELIGIBILITY:
Inclusion Criteria:- AMI developed < 12-hr - Reference lumen diameter (RLD) of infarct related artery (IRA) > 3.0 mmExclusion criteria:- electrical instability- patient is in Killip class 3 or 4 of heart failure- implanted electronic devices are present- all implants held by magnets/fragments/devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-04; Study Completion 2005-12

PRIMARY OUTCOMES:
MRI assessment of LV volumes during hospitalisation and after 3 months

SECONDARY OUTCOMES:
ST-resolution after PCI, serial cardiac enzymes, myocardial blush grade, TIMI flow rate

CONTACTS AND LOCATIONS:
Overall Officials: B. Rensing, MD, PhD, Study Chair — St. Antonius Hospital
Locations (1):
- St Antonius Hospital, Nieuwegein, Netherlands